CLINICAL TRIAL: NCT04190251
Title: PANDIA IRIS: Patients With Diabetes and Kidney Failure, an Interdisciplinary Medication Adherence Support Program
Acronym: PANDIA_IRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Collaborators: pharmaSuisse (Unknown); santésuisse (Unknown); Curafutura (Unknown)
Responsible Party: Principal Investigator, Marie Schneider, Pr. Schneider Marie P., PhD, Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PB_2016-01674(454/15)
Record Dates: First submitted 2019-10-22; First posted 2019-12-09 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic
Keywords: Medication adherence; Diabetes Mellitus; Renal Insufficiency, Chronic; Interprofessional Relations
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Medication Adherence; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group A (Other): Intervention group A will benefit of the medication adherence support program during 12 months. Adherence will be monitored using an Electronic Monitoring system (EM, named MEMS®; Aardex Ltd.) during 24 months. At each pharmacy visits, the pharmacist will conduct an 15 minutes, semi-structured interview based on Fisher's sociocognitiv model with the patients. A summary and the adherence graph will be send to all the involved health professionals
  Interventions: Other: Inteprofessional medication adherence support program (IMAP)
- Intervention group B (Other): Intervention group A will benefit of the medication adherence support program during 6 months. Adherence will be monitored using an Electronic Monitoring system (EM, named MEMS®; Aardex Ltd.) during 24 months. At each pharmacy visits, the pharmacist will conduct an 15 minutes, semi-structured interview based on Fisher's sociocognitiv model with the patients. A summary and the adherence graph will be send to all the involved health professionals
  Interventions: Other: Inteprofessional medication adherence support program (IMAP)

INTERVENTIONS:
Other: Inteprofessional medication adherence support program (IMAP) — In addition to usual care, patients participate in a medication adherence support program combining an Electronic Monitoring system (EM, named MEMS®; Aardex Ltd) and motivational semi-structured interviews. This programm is done by the Unisanté's community pharmacists, in coordination with medical and nurse staff , to support medication adherence and to promote continuity of care. The intervention is held at the Unisanté's community pharmacy. For patients not speaking french, english, or italien, the interviews will be done with a interpreter.

SUMMARY:
Monocentric, randomised, controlled and open study. Subjects will be included prospectively and consecutively and randomly assigned into two groups. Intervention group A will benefit a medication adherence support program during 12 months while intervention group B during 6 months only. Adherence will be monitored using an Electronic Monitoring system (EM, named MEMS®; Aardex Ltd.) during 24 months. At each pharmacy visit, the pharmacist will conduct a semi-structured interview in 15 minutes based on Fisher's sociocognitive model with the patients. A summary of the interview and the adherence graph will be send to the patient' health professionals.

DETAILED DESCRIPTION:
In addition to usual care, patients are included in a medication adherence support program combining an Electronic Monitoring system (EM, named MEMS®; Aardex Ltd) and motivational semi-structured interviews. This programm is held by the Unisanté's community pharmacists*, in coordination with medical and nurse staff , to support medication adherence and to promote the continuity of care. For patients not speaking french, english, or italian, the interviews will be done with a interpreter.

The medication adherence data will be analysed in both groups along with clinical data obtained through draw samples regularly prescribed by the physician.

*Since the 1st January 2019, the Policlinique Médicale Universitaire became Unisanté, University Center for Primary Care and Public Health (Lausanne, Switzerland).

ELIGIBILITY:
Inclusion criteria:

* MDRD or CKD-EPI eGFR ≤60 ml/min/1.73m2 or albumin/creatinin >30mg/mmol
* Type 2 diabetes
* At least one medication in the following list : oral antidiabetics and/or statins and/or antihypertensive drugs and/or aspirin
* Patients speaking french, english or italian or interpreter present at each pharmacy visit
* Patients have to sign the written consent form
* Patients have to agree to use the Electronic Monitoring system (EM, named MEMS®; Aardex Ltd)
* Complete laboratory exams in the last 6 months: eGFR and HbA1c and (albumin/creatinin ratio or total cholesterol + LDL + HDL)

Exclusion Criteria:

* Not being able to understand or sign the consent form
* Pregnancy
* Recent cancer diagnosis
* Cognitive disorder
* The subject does not manage the treatment alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Medication adherence (longitudinal data) | 24 months
  Implementation and persistance during the intervention phase (6 or 12 months) and during the post-intervention phase (18 months or 12 months)

SECONDARY OUTCOMES:
Clinical outcomes | Baseline, 6 monts and 12 months post-intervention
  ADVANCE kidney score
Clinical outcomes | Baseline, 6 monts and 12 months post-intervention
  UKPDS score
Medication adherence | 6 months or 12 months post-intervention phase
  Number of patients with an electronic medication adherence ≤ 30% for at least one medication throughout two successive pharmacy visits during the post-intervention phase
Patients' satisfaction | At 6 months or 12 months (end of the intervention phase) or at the stop of the study (24 months if the patient ends the study or between the end of the intervention phase (6 months or 12 months) and 24 months.
  In depths and semi-structured interviews to assess patient's opinions about the program

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Paule Schneider, Prof., Principal Investigator — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland; Carole Bandiera, PhD student, Principal Investigator — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland; Anne Zanchi, PhD-PD, Principal Investigator — CHUV (Centre hospitalier Universitaire Vaudois)
Locations (2):
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - Unisante, Lausanne, Canton of Vaud

REFERENCES:
- [Derived] Bandiera C, Dotta-Celio J, Locatelli I, Nobre D, Wuerzner G, Pruijm M, Lamine F, Burnier M, Zanchi A, Schneider MP. The differential impact of a 6-versus 12-month pharmacist-led interprofessional medication adherence program on medication adherence in patients with diabetic kidney disease: the randomized PANDIA-IRIS study. Front Pharmacol. 2024 Jan 24;15:1294436. doi: 10.3389/fphar.2024.1294436. eCollection 2024. PMID 38327981
- [Derived] Bandiera C, Lam L, Locatelli I, Dotta-Celio J, Duarte D, Wuerzner G, Pruijm M, Zanchi A, Schneider MP. Understanding reasons and factors for participation and non-participation to a medication adherence program for patients with diabetic kidney disease in Switzerland: a mixed methods study. Diabetol Metab Syndr. 2022 Sep 27;14(1):140. doi: 10.1186/s13098-022-00898-7. PMID 36167584
- [Derived] Bandiera C, Dotta-Celio J, Locatelli I, Nobre D, Wuerzner G, Pruijm M, Lamine F, Burnier M, Zanchi A, Schneider MP. Interprofessional Medication Adherence Program for Patients With Diabetic Kidney Disease: Protocol for a Randomized Controlled and Qualitative Study (PANDIA-IRIS). JMIR Res Protoc. 2021 Mar 19;10(3):e25966. doi: 10.2196/25966. PMID 33739292